# Statistical Analysis Plan (SAP)

A Phase II, Placebo-Controlled, Randomized, Double-Blind Study to Assess the Safety, Tolerability and Efficacy of terpenes-enriched CBD-predominant cannabis oil, Administered to Pediatric Subjects with Autism Spectrum Disorder (ASD)

Trial Registration: ClinicalTrials.gov Identifier: NCT07199218

SAP Version: Version 1.0; September 01, 2025

Protocol No.: 0336-24-SZMC

Protocol Reference: Protocol Version 3.0, September 1, 2025.

### **SAP** revision history

| Version | Author | Date | Description |
|---------|--------|------|-------------|

| Approvals: | |
|-----------------------------------------|--------------------|
| | Date and signature |
| Drafted by Dr. Nardine Fahoum – Khalefa | |
| Statistician | |
| Bazelet Group (Or Akiva, Israel) | |
| Reviewed by Dr. Noa Raz | |
| chief scientist | |
| Bazelet Group (Or Akiva, Israel) | |
| Approved by Principal Investigator: | |
| Prof. Adi Aran | |
| Shaare Zedek Medical Center | |

## 1 Introduction

## 1.1 Background and rationale

Autism spectrum disorder (ASD) encompasses a wide range of neurodevelopmental disorders with diverse etiologies and symptoms. Efforts to develop a single pharmacological treatment for the core symptoms of ASD have been unsuccessful.¹ Approved antipsychotic medications for managing associated irritability often result in substantial metabolic side effects. <sup>2,3</sup> Cannabidiol (CBD), a non-psychoactive cannabinoid, targets multiple neuronal and glial pathways to reduce excitation and inflammation.<sup>4-11</sup>,<sup>12-15</sup> In contrast, tetrahydrocannabinol (THC), a psychoactive cannabinoid, directly activates the endocannabinoid system, which is impaired in ASD, and decreases social anxiety and hostility. <sup>16</sup> Preliminary trials in children with ASD have demonstrated the efficacy of a CBD-predominant formulation combined with low-dose THC.<sup>17</sup> Preclinical data suggest that efficacy may be further enhanced by enriching cannabinoid compounds with selected terpenes, which activate CB1 and CB2 receptors both directly and by modulating THC interactions at these receptors.<sup>18-23</sup>

The present study is designed to assess the combined impact of CBD, terpenes, and low-dose THC. We hypothesize that this combination will lead to significantly greater improvements in disruptive behaviors and core autistic symptoms compared with placebo.

## 1.2 Objectives

The primary aim is to assess the effect of the study drug compared to placebo on behavioral problems, using the Aberrant Behavior Checklist-Irritability Subscale (ABC-I) score - change from baseline to week 8.

The main secondary aim is to assess the effect of the study drug compared to placebo on core ASD symptoms using the Vineland ™ Adaptive Behavior Scales (3rd edition, VABS3)-Socialization Domain Score, and the Social Responsiveness Scale 2nd edition (SRS-II) total score - change from baseline to week 8.

Other secondary aims include: (1) To assess the tolerability and safety of the study drug compared to placebo, using detailed questionnaires, physical examination, blood count, and liver enzyme tests. (2) To assess global change in ASD-associated symptoms using the Clinical Global Impression- Improvement (CGI-I) and the Caregiver Global Impression of Change (CGIC) assessments – change from baseline to week 8. (3) To assess changes in the quality of life, sleep parameters, and gastrointestinal problems using the Pediatric Quality of Life Inventory (PedsQL), the Quality of Life in Autism Questionnaire (QOLA) – Parent version, the Children's Sleep Habits Questionnaire (CSHQ) and a modified gastrointestinal sign and symptoms inventory (GISSI) - change from baseline to week 8. (4) To compare the effect of CBD-predominant, terpene-enriched cannabis oil (study drug) and terpenes-enriched CBD oil, using the above assessments - change from baseline to week 8 and week 17.

## 2 Study Methods

## 2.1 Trial design

This is a phase II, randomized, double-blind, placebo-controlled, parallel-group study, involving 78 children with ASD and behavioral problems, age 4-12 years. Participants who will pass screening will be randomized (in a 1:1 ratio) to receive either placebo or terpenes-enriched

CBD-predominant cannabis oil (CBD: 3.6 mg/kg twice daily, terpenes: 0.25mg/kg twice daily, and THC: 0.128 mg/kg twice daily). The treatment will be given orally as an add-on to any existing treatment, for 8 weeks. The treatment dose will be up-titrated over 8 days.

After completing the first 8-week period, participants who received placebo will receive pure CBD (3.8 mg mg/kg twice daily) enriched with terpenes (0.25mg/kg twice daily), and participants who received the study drug will continue with the same treatment for another 8 weeks of the second phase.

### 2.2 Randomization

A randomization scheme will be generated by an external unblinded biostatistician. The blocked randomization will be performed using SAS statistical software V9.4 via the plan procedure with a fixed block size. The randomization scheme and lists will be sent to the study site. The randomization list will include sequential numbers and assigned 4-letter codes. Randomization will be kept at a 1:1 ratio. The randomization list will be encrypted by password and will be sent prior to first dosing to the principal investigator.

## 2.3 Sample Size

The planned sample size is 78 participants (39 per arm). This calculation, including assumptions about expected effect size and dropout rate, is described in detail in Protocol 0336-24-SZMC, Section 13 (Statistical Considerations).

### 2.4 Framework

This trial is designed as a **superiority trial**. The primary hypothesis is that terpene-enriched CBD-predominant cannabis oil will be superior to placebo in reducing irritability symptoms in children with ASD, as measured by change in ABC-I score from baseline to week 8.

## 2.5 Statistical interim analysis and stopping guidance

This study incorporates an adaptive design with interim analysis by an external, non-blinded biostatistician. Final sample size will be determined based on that interim analysis

An independent Data and Safety Monitoring Board (DSMB) will review the interim analyses as needed, although no formal stopping rules are defined for this study, and will ensure that all trial data remain confidential.

## 2.6 Timing of Analyses

The final statistical analysis will be conducted after completion of follow-up for the last randomized participant, once all data through week 17 have been collected.

## 2.7 Timing of outcome assessments

On-site visits: 5 visits: Screening (visit #1), Baseline (visit #2), 4 weeks (visit #3), 8 weeks (visit #4 - end of the first phase) and 17 weeks (visit #5 - end of the second phase). Phone visits to document compliance and adverse events: Three visits at study onset- (days 4, 8, and 12) and another 3 visits on weeks 6, 11, and 13.

## 3 Statistical Principals

### 3.1 Confidence intervals and P values

Hypothesis testing, unless otherwise indicated, will be 2-sided and performed at the 5% significance level. When confidence intervals (CI) are presented, they will be 2-sided with a confidence coefficient of 95%.

No adjustments for multiplicity will be made for the secondary efficacy analyses in this study. Nominal p-values will be presented for informational purposes only.

### 3.2 Adherence and Protocol deviations

### 3.2.1 Adherence

Adherence is defined as the proportion of study doses actually taken during the randomized phase (Days 1–56). Adherence will be assessed from caregiver reports collected at prespecified phone/Zoom visits (Days 4, 8, 12,42) and at on-site visits.

Overall duration of exposure in days will be computed for each randomized subject using the following equation:

End date of study treatment - start date of study treatment +1

Summary statistics for treatment compliance will be displayed by arm (n, mean, median, standard deviation, minimum, and maximum).

### 3.2.2 Deviations from the Protocol

Neither the Principal Investigator nor any sub-investigator is authorized to deviate from the protocol, except as permitted under section 4.5.4(b) of ISO 14155:2011 and 21 CFR 812.150(a)(4). Specifically, protocol deviations may only be made or reported if they affect a subject's rights, safety, or well-being, or the scientific integrity of the clinical investigation.

Under emergency circumstances, deviations from the protocol to protect the rights, safety, and well-being of human subjects may proceed without prior approval of the sponsor and the EC/IRB/Helsinki Committee. Such deviations shall be documented and reported to the sponsor and the EC/IRB/Helsinki Committee as soon as possible.

The research coordinator will prepare the EC/IRB /Helsinki Committee Notifications letter using the EC Notification Form if any reportable serious deviations or adverse events were recorded and send them to the Ethics Committee/Institutional Review Board/Helsinki Committee and Principal Investigator, according to this protocol.

All notifications will be carried out within the time frames specified by local regulatory authorities.

## 3.3 Analysis populations

### 3.3.1 Safety Population

The Safety population is defined as all enrolled subjects who received at least one dose of study medication (including placebo). Safety analyses will be performed using the Safety population and subjects will be analyzed according to the treatment received in each part.

### 3.3.2 Intent to Treat Population (ITT)

ITT population will include all randomized subjects regardless of receiving study drug or being assessed in study measurements.

If all randomized subjects receive at least one dose of study drug, the ITT population and the safety population will be equal, and will be reported as one.

### 3.3.3 Per Protocol Population (PP)

The PP population will include all randomized subjects who completed the study according to protocol.

The primary efficacy analysis will be conducted on the intention-to-treat (ITT) population, defined as all randomized participants analysed according to their assigned treatment arm, regardless of adherence or protocol deviations. A supportive secondary analysis will be performed on the per-protocol (PP) population, consisting of participants who complete the study without major protocol deviations, in order to assess the robustness and consistency of the results.

## **4 Trial Population**

## 4.1 Screening data and Eligibility

Screening will occur at Visit 1 (Day -90 to Day -1). Eligibility assessments include DSM-5 diagnostic confirmation with CARS-2, CGI-S, ABC-I, SRS-II, medical history, vitals/exam, and labs, as outlined in the protocol schedule of activities. We will report screening data to describe the representativeness of the randomized cohort as follows:

- **CONSORT-style flow:** numbers screened, eligible, consented, randomized, and not randomized, with reasons for screen failure.
- Reasons for screen failure (tabulated counts and %): did not meet inclusion
  thresholds (e.g., ABC-I <18, SRS-II <66, CGI-S <4, age/weight out of range), met exclusion
  criteria (e.g., recent seizures/antiepileptic change, recent cannabinoid use, clinically
  significant abnormal labs, prohibited comedications), declined consent, logistical
  reasons.</li>
- **Descriptive comparison**: age and sex distributions in screened vs randomized participants, to comment on representativeness.

Eligibility criteria (full detail in **Protocol 0336-24-SZMC**) are summarized here for analysis clarity.

#### **Inclusion criteria**

Age 4–12 years.

- ASD diagnosis per DSM-5, confirmed by CARS-2.
- CGI-S ≥4 (moderate or greater severity).
- ABC-I ≥18.
- SRS-II total T ≥66.

#### **Exclusion criteria**

- Weight <12.5 kg or  $\geq$ 57.5 kg.
- Current/past heart failure, drug addiction, schizophrenia/psychosis/bipolar/PTSD/MDD, or schizophrenia in a first-degree relative.
- Seizure or change in antiepileptic medication in the 4 months before randomization.
- Clinically significant abnormal physical exam or labs (e.g., heart, liver, renal function).
- Change in pharmacologic/behavioral treatment or home/school setting within 4 weeks prior to randomization, or planned changes during the study.
- Cannabinoid treatment within 4 weeks prior to randomization.
- Predicted low compliance with study procedures.
- Concurrent opiates or alcohol use.

## 4.2 Withdrawal/Follow-up

Withdrawal will be classified at four levels:

- 1. **From intervention** participant discontinues study drug (reasons will be documented)
- 2. **From follow-up** participant stops attending visits/assessments (lost to follow-up)
- 3. **Withdrawal of consent** participant/caregiver withdraws consent for further participation (reasons will be documented)
- 4. **Protocol-mandated discontinuation** Investigator/sponsor stops intervention and/or follow-up (e.g., safety reasons, ineligibility discovered later).

Withdrawal status (and reason, if provided) will be captured at the time of discontinuation and/or at the next scheduled contact (phone/Zoom or on-site), using the visit schedule and windows defined in the protocol. Compliance and adverse events are collected repeatedly at these visits, enabling precise dating of discontinuation and last contact.

Reasons will be recorded and coded into prespecified categories: adverse event/tolerability, lack of efficacy, caregiver decision/burden, non-adherence, intercurrent illness/procedure, protocol-specified ineligibility discovered post-randomization, logistical/administrative, and other.

Presentation will include:

• **CONSORT flow**: numbers screened, randomized, treated, completed, withdrawn (by level and reason), and analysed.

• Tables by treatment arm: counts (%) for each withdrawal level (intervention only; follow-up; consent withdrawal), timing and reason category.

## 4.3 Baseline patient characteristics

Demographics variables and baseline characteristics will be summarized for the Safety population. Demographic and baseline data will be presented overall and by treatment sequence.

Demographic variables include age, sex, ethnicity, height, weight, and body mass index (BMI) collected at the Screening Visit.

Baseline characteristics include the following:

- DSM-5 levels of support required
- CARS-2
- VABS-3
- CGI-S,
- ABC-I
- SRS
- NVIQ
- Etiological factors
- Comorbidities
- History of autistic regression
- Diet
- Behavioural treatments
- Impact of high fever on social deficits status
- Concomitant medications

Data from continuous variables will be tested for normal distribution. Summaries of continuous variables that are normally distributed will be presented as means and standard deviations or medians and inter quartiles for skewed data. Categorical variables will be presented as frequencies and percentages.

## 5 Analysis

### 5.1 Outcomes

#### **Primary endpoint**

<u>ABC-I</u>: The ABC<sup>24,25</sup> is a caregiver-completed questionnaire with 58 items, organized into five subscales. The ABC-I (irritability) subscale consists of 15 items that measure the emotional and behavioral symptoms of ASD, including aggression toward others, deliberate self-injuriousness,

temper tantrums, depressed mood and rapidly changing moods. The ABC-I has been accepted as the gold standard for measuring irritability in medication trials for  $ASD^{26}$  and therefore, we will use it as the primary endpoint in this study. Individual items are rated from 0 (never a problem) to 3 (severe problem) and the ABC-I total is the sum of the 15 items (range 0–45; higher = worse).

Assessed at baseline, Week 4, Week 8, and Week 17; the primary endpoint is the change in ABC-I from baseline to Week 8.

#### Main secondary outcome measures

<u>VABS-III</u> <sup>27</sup>: The VABS is a semi-structured caregiver interview designed to assess functional skills in three domains: Communication, Socialization, and Daily Living Skills. It also contains a short Maladaptive Behavior Domain. The Adaptive Composite Score estimates overall adaptive behavior. Vineland items are scored based on an open-ended question as 0 (behavior not performed), 1 (performed sometimes), or 2 (performed on a regular basis). The instrument provides Standard scores (mean = 100, SD = 15) and Age Equivalent scores.

Assessed at baseline and Week 8; analysed as change from baseline to Week 8.

SRS (Hebrew version) <sup>28,29</sup>: this 65-item caregiver or teacher questionnaire contains five subscales: Social Awareness, Social Cognition, Social Communication, Social Motivation, and Autistic Mannerisms, which respectively measure the ability to recognize social cues, the ability to interpret social cues, the ability to use expressive verbal and nonverbal language skills, the ability to engage in social-interpersonal behaviors, and the tendency to display stereotypical behaviors and restricted interests characteristic of autism. Each item is rated on a four-point Likert scale, (0 to 3, total scores range from 0 to 195) with a higher score indicating greater impairment. Each subscale can be converted into T-score. The SRS Total T-score reflects the sum of the T-scores for the five scales. SRS T-scores between 60 and 75 indicate a mild to moderate social impairment whereas scores above 75 indicate a "severe" level. The caregivers will complete the SRS based on the participant's behavior over the previous 6 weeks. The SRS has been used extensively to assess behavioral problems in ASD research <sup>30-35</sup>

Assessed at baseline, Week 4, Week 8, and Week 171; analysed as change from baseline to Week 8.

### Other secondary outcome measures:

<u>CGI-I</u>: The CGI <sup>36</sup> is a 7-point scale designed to measure the severity of illness (CGI-S) and, an overall improvement from baseline (CGI-I). This measure has been used in many clinical trials in ASD.<sup>37-39</sup> Scores in the severity scale range from 1 (normal) through to 7 (amongst the most severely ill patients); in the improvement scale, scores range from 1 (very much improved) through 4 (unchanged) to 7 (very much worse).

*CaGIC*: this is a 7-point scale designed to measure the overall improvement from baseline. This measure is completed by the primary caregivers and is similar to the CGI-I

<u>Autism Impact Measure (AIM)</u><sup>40,41</sup>: This is a 41-item caregiver-reported questionnaire designed to characterize core symptoms of ASD in individuals aged 3–18 years

<u>Multidimensional Assessment of Preschool Disruptive Behavior (MAP-DB)</u><sup>42</sup>: This 40-item caregiver-reported questionnaire assesses behavior across four domains: Temper Loss, Noncompliance, Aggression, and Low Concern for Others. It is available in three age-specific versions: 3-5 years, 6-8 years, and 9-10+ years.

<u>Emotion dysregulation inventory (EDI)</u><sup>43</sup>: This 30-item caregiver-reported questionnaire assesses observable signs of poor emotion regulation in children with autism.

<u>Behavior Rating Inventory of Executive Function (BRIEF)</u><sup>44</sup>: this is an 88 items Hebrew validated questionnaire, consists of 8 subscales, grouped into two index scores—Behavioral Regulation Index and Metacognition Index. Raw scores are converted into age- and sex-normed T scores.

Children's Sleep Habits Questionnaire (CSHQ)<sup>45</sup>: this is a 33 items Hebrew validated questionnaire. A higher score reflects more significant sleep disturbances (range: 33–99, a score of ≥41 classifies a "poor sleeper). The CSHQ has eight subscales: bedtime resistance; sleep onset delay; sleep duration; sleep anxiety; night waking; parasomnias; sleep-disordered breathing; and daytime sleepiness. This questionnaire has been used extensively in previous research in ASD

<u>Pediatric Quality of Life Inventory (PedsQL)</u><sup>46</sup>: The PedsQL™ is a validated tool for measuring health-related quality of life (HRQOL) in children aged 2–18 years with acute or chronic health conditions, as well as in healthy individuals. Different formats exist, including parent proxy reports and age-specific versions, which use identical items with age-appropriate language. This study will use the parent proxy report of the PedsQL 4.0 Generic Core Scales, which assess physical, mental, social health, and role functioning.

Quality of Life in Autism Questionnaire (QOLA) – Parent version: <sup>47</sup>The QOLA is a 48-item tool with two subscales to measure quality of life in parents of children with ASD. Part A (QoL subscale) includes 28 items assessing parents' overall quality of life, with scores ranging from 28 to 140 (higher scores indicate greater QoL). Part B (impact of ASD symptoms subscale) includes 20 items evaluating how problematic a child's ASD-related difficulties are for the parent, with scores ranging from 20 to 100 (higher scores indicate fewer problems).

<u>Modified gastrointestinal signs and symptoms inventory (GISSI)</u>: This 15-item questionnaire was adapted to this study based on the GISSI-17,<sup>48</sup> a brief parent-report screen for common gastrointestinal problems in children with ASD.

Blood samples- (15 ml) will be collected at 0 and 8 weeks.

- Complete blood count (CBC), liver transaminases (LTs) and total bilirubin will be measured as part of the safety analyses.
- Plasma levels of 7-carboxy-CBD<sup>49</sup> will be assessed to determine individual bioavailability of CBD. At 2-month, blood will be collected 3-4 hours post treatment administration.
- Serum endocannabinoids (ECs)<sup>50,51</sup> and relative mRNA expression levels (real-time PCR) of components of the eCB system in whole blood,<sup>51</sup> RNA-sequencing of whole blood samples (transcriptome),<sup>52</sup> and plasma proteome,<sup>53</sup> will be assessed to explore possible markers of treatment response.

Stool samples will be collected at 0 and 8 weeks.

 Gut microbiota was demonstrated to be associated with ASD as well as symptom severity in multiple studies.<sup>54-56</sup>

Assessment of the other secondary outcomes is detailed within the protocol

### 5.2 Statistical Methods

The primary endpoint, change in ABC-I from baseline to Week 8, will be analysed under a superiority framework using a mixed model for repeated measures (MMRM). The model will include fixed effects for treatment (study drug vs placebo), visit (Baseline, Week 4, and Week 8), and the treatment-by-visit interaction, with a subject-level random effect. The primary contrast is the adjusted difference between arms at Week 8, reported as a least-squares (LS) mean difference with two-sided 95% confidence interval and p-value.

Secondary analyses will be conducted using the same methodology as for the primary ABC-I endpoint.

Sensitivity analyses will include per-protocol analysis and may utilize multiple imputation to confirm the robustness of findings.

The primary report will focus on odds ratios (OR) and 95% confidence intervals (CI). Additionally, a secondary analysis will evaluate the proportion of participants achieving the minimal clinically important difference (MCID) using a chi-square test or logistic regression analysis to compare proportions between groups. The analysis of the Vineland Adaptive Behavior Scales, Third Edition (VABS-III), will utilize Growth Scale Values (GSV), with adjustments for participants transitioning between age categories during the study.

Data from continuous variables will be tested for normal distribution. Summaries of continuous variables that are normally distributed will be presented as means and standard deviations or medians and inter quartiles for skewed data. Categorical variables will be presented as frequencies and percentages. If distributions are not normal, rank-based approaches will be applied.

## 5.3 Missing data

The primary analyses will use mixed models for repeated measures, which incorporate all available observations under a missing at random (MAR) assumption and do not require single imputation. The primary analysis assumes that ABC-I scores are MAR, an assumption deemed reasonable for this study. Missing data are unlikely to differ systematically from observed values for unknown reasons. We will describe the extent and timing of missing data by arm and visit, including numbers and percentages missing for each endpoint and known reasons. To assess robustness to departures from MAR, we will perform multiple imputation as a sensitivity analysis.

### 5.4 Harms

All subjects who enter the study will be assessed for safety. Safety will be monitored by structured monthly parental reports, immediate intercurrent reports of exceptional phenomena, physical examination, detailed interview, and adverse event (AE) assessment at each visit.

### 5.4.1 Adverse Events

AEs will be monitored using a 31-item modification of the Dosage Record and Treatment Emergent Symptom Scale. Recent health concerns, use of medical services, and changes in study treatment dose and concomitant medications will be recorded. BMI, pulse rate, and blood pressure will be assessed at each clinic visit. New AEs or worsening of previously reported AEs will be rated **mild** (present but not persistent or requiring intervention), **moderate** (requiring intervention), or **severe** (posing a severe problem and requiring immediate intervention); hospitalization will be documented as a serious adverse event. The Principal Investigator will evaluate all AEs for timing, biological plausibility, alternative causes, dose–response relationship, and prior knowledge to determine relatedness to the study drug as not related, unlikely, possibly, probably, or definitely related. AEs will be reported and managed according to 21 CFR (§812.150(a)(1), §812.46(b), §812.150(b)(1)), MEDDEV 2.7/3 (Dec 2010), and ICH-GCP guidelines. Anticipated AEs include rare insomnia, irritability, and intolerance of the taste and smell. An overview of the incidence and frequency of AEs will be presented by treatment condition in the Safety population.

### **5.4.2 Blood samples**

Complete blood count, liver transaminases and total bilirubin will be measured as part of the safety analyses.

### 5.5 Statistical software

SAS (PROC MIXED), R (lme4 package), or equivalent statistical software.

## 6 References

- 1. Lord C, Elsabbagh M, Baird G, Veenstra-Vanderweele J. Autism spectrum disorder. *Lancet*. Aug 11 2018;392(10146):508-520. doi:10.1016/s0140-6736(18)31129-2
- 2. Scahill L, Jeon S, Boorin SJ, et al. Weight Gain and Metabolic Consequences of Risperidone in Young Children With Autism Spectrum Disorder. *J Am Acad Child Adolesc Psychiatry*. May 2016;55(5):415-23. doi:10.1016/j.jaac.2016.02.016
- 3. Goel R, Hong JS, Findling RL, Ji NY. An update on pharmacotherapy of autism spectrum disorder in children and adolescents. *Int Rev Psychiatry*. Feb 2018;30(1):78-95. doi:10.1080/09540261.2018.1458706
- 4. Atalay S, Jarocka-Karpowicz I, Skrzydlewska E. Antioxidative and Anti-Inflammatory Properties of Cannabidiol. *Antioxidants (Basel)*. Dec 25 2019;9(1)doi:10.3390/antiox9010021
- 5. Ribeiro A, Ferraz-de-Paula V, Pinheiro ML, et al. Cannabidiol, a non-psychotropic plant-derived cannabinoid, decreases inflammation in a murine model of acute lung injury: role for the adenosine A(2A) receptor. *Eur J Pharmacol*. Mar 5 2012;678(1-3):78-85. doi:10.1016/j.ejphar.2011.12.043
- 6. Furgiuele A, Cosentino M, Ferrari M, Marino F. Immunomodulatory Potential of Cannabidiol in Multiple Sclerosis: a Systematic Review. *J Neuroimmune Pharmacol*. Jan 25 2021:1-19. doi:10.1007/s11481-021-09982-7
- 7. Kozela E, Lev N, Kaushansky N, et al. Cannabidiol inhibits pathogenic T cells, decreases spinal microglial activation and ameliorates multiple sclerosis-like disease in C57BL/6 mice. *Br J Pharmacol*. Aug 2011;163(7):1507-19. doi:10.1111/j.1476-5381.2011.01379.x

- 8. Kozela E, Juknat A, Kaushansky N, Rimmerman N, Ben-Nun A, Vogel Z. Cannabinoids decrease the th17 inflammatory autoimmune phenotype. *J Neuroimmune Pharmacol*. Dec 2013;8(5):1265-76. doi:10.1007/s11481-013-9493-1
- 9. Kozela E, Juknat A, Gao F, Kaushansky N, Coppola G, Vogel Z. Pathways and gene networks mediating the regulatory effects of cannabidiol, a nonpsychoactive cannabinoid, in autoimmune T cells. *J Neuroinflammation*. Jun 3 2016;13(1):136. doi:10.1186/s12974-016-0603-x
- 10. Burstein S. Cannabidiol (CBD) and its analogs: a review of their effects on inflammation. *Bioorg Med Chem.* Apr 1 2015;23(7):1377-85. doi:10.1016/j.bmc.2015.01.059
- 11. Mecha M, Feliú A, Iñigo PM, Mestre L, Carrillo-Salinas FJ, Guaza C. Cannabidiol provides long-lasting protection against the deleterious effects of inflammation in a viral model of multiple sclerosis: a role for A2A receptors. *Neurobiol Dis.* Nov 2013;59:141-50. doi:10.1016/j.nbd.2013.06.016
- 12. Kozela E, Pietr M, Juknat A, Rimmerman N, Levy R, Vogel Z. Cannabinoids Delta(9)-tetrahydrocannabinol and cannabidiol differentially inhibit the lipopolysaccharide-activated NF-kappaB and interferon-beta/STAT proinflammatory pathways in BV-2 microglial cells. *J Biol Chem.* Jan 15 2010;285(3):1616-26. doi:10.1074/jbc.M109.069294
- 13. Juknat A, Pietr M, Kozela E, et al. Differential transcriptional profiles mediated by exposure to the cannabinoids cannabidiol and  $\Delta 9$ -tetrahydrocannabinol in BV-2 microglial cells. *Br J Pharmacol*. Apr 2012;165(8):2512-28. doi:10.1111/j.1476-5381.2011.01461.x
- 14. Juknat A, Pietr M, Kozela E, et al. Microarray and pathway analysis reveal distinct mechanisms underlying cannabinoid-mediated modulation of LPS-induced activation of BV-2 microglial cells. *PLoS One*. 2013;8(4):e61462. doi:10.1371/journal.pone.0061462
- 15. Juknat A, Gao F, Coppola G, Vogel Z, Kozela E. miRNA expression profiles and molecular networks in resting and LPS-activated BV-2 microglia-Effect of cannabinoids. *PLoS One.* 2019;14(2):e0212039. doi:10.1371/journal.pone.0212039
- 16. Szkudlarek HJ, Desai SJ, Renard J, et al. Delta-9-Tetrahydrocannabinol and Cannabidiol produce dissociable effects on prefrontal cortical executive function and regulation of affective behaviors. *Neuropsychopharmacology*. Mar 2019;44(4):817-825. doi:10.1038/s41386-018-0282-7
- 17. Aran A, Harel M, Cassuto H, et al. Cannabinoid treatment for autism: a proof-of-concept randomized trial. *Mol Autism*. Feb 3 2021;12(1):6. doi:10.1186/s13229-021-00420-2
- 18. Raz N, Eyal AM, Davidson EM. Optimal Treatment with Cannabis Extracts Formulations Is Gained via Knowledge of Their Terpene Content and via Enrichment with Specifically Selected Monoterpenes and Monoterpenoids. *Molecules*. Oct 15 2022;27(20)doi:10.3390/molecules27206920
- 19. Staben J, Koch M, Reid K, et al. Cannabidiol and cannabis-inspired terpene blends have acute prosocial effects in the BTBR mouse model of autism spectrum disorder. *Front Neurosci.* 2023;17:1185737. doi:10.3389/fnins.2023.1185737
- 20. Raz N, Eyal AM, Zeitouni DB, et al. Selected cannabis terpenes synergize with THC to produce increased CB1 receptor activation. *Biochem Pharmacol*. Jun 2023;212:115548. doi:10.1016/j.bcp.2023.115548
- 21. Câmara JS, Perestrelo R, Ferreira R, Berenguer CV, Pereira JAM, Castilho PC. Plant-Derived Terpenoids: A Plethora of Bioactive Compounds with Several Health Functions and Industrial Applications-A Comprehensive Overview. *Molecules*. Aug 15 2024;29(16)doi:10.3390/molecules29163861
- 22. Rava A, Buzzelli V, Feo A, et al. Role of peroxisome proliferator-activated receptors  $\alpha$  and  $\gamma$  in mediating the beneficial effects of  $\beta$ -caryophyllene in a rat model of fragile X syndrome. *Prog Neuropsychopharmacol Biol Psychiatry*. Jan 10 2025;136:111234. doi:10.1016/i.pnpbp.2024.111234
- 23. Alayoubi M, Rodrigues A, Wu C, et al. Elucidating interplay between myrcene and cannabinoid receptor 1 receptors to produce antinociception in mouse models of neuropathic pain. *Pain*. Mar 18 2025;doi:10.1097/j.pain.0000000000003558

- 24. Aman MG, Singh NN, Stewart AW, Field CJ. The aberrant behavior checklist: a behavior rating scale for the assessment of treatment effects. *American journal of mental deficiency*. Mar 1985;89(5):485-91.
- 25. Aman M. Aberrant behaviour checklist—community. East Aurora, NY: Slosson Educational Publications; 1994.
- 26. Fung LK, Mahajan R, Nozzolillo A, et al. Pharmacologic Treatment of Severe Irritability and Problem Behaviors in Autism: A Systematic Review and Meta-analysis. *Pediatrics*. Feb 2016;137 Suppl 2:S124-35. doi:10.1542/peds.2015-2851K
- 27. Taylor J, Watkins C, Kaplin A. Kleine-Levin syndrome: a disease in its own right? *Nat Clin Pract Neurol*. Oct 2008;4(10):534-5. doi:ncpneuro0900 [pii]

### 10.1038/ncpneuro0900 [doi]

- 28. Constantino JN, Gruber CP. The Social Responsiveness Scale (SRS) (Manual). Los Angeles: Western Psychological Services. 2005;
- 29. Ben-Sasson A, Lamash L, Gal E. To enforce or not to enforce? The use of collaborative interfaces to promote social skills in children with high functioning autism spectrum disorder. *Autism: the international journal of research and practice*. Sep 2013;17(5):608-22. doi:10.1177/1362361312451526
- 30. Aman MG, Findling RL, Hardan AY, et al. Safety and Efficacy of Memantine in Children with Autism: Randomized, Placebo-Controlled Study and Open-Label Extension. *Journal of child and adolescent psychopharmacology*. Mar 15 2016;doi:10.1089/cap.2015.0146
- 31. Freitag CM, Jensen K, Elsuni L, et al. Group-based cognitive behavioural psychotherapy for children and adolescents with ASD: the randomized, multicentre, controlled SOSTA net trial. *Journal of child psychology and psychiatry, and allied disciplines*. May 2016;57(5):596-605. doi:10.1111/jcpp.12509
- 32. Minshawi NF, Wink LK, Shaffer R, et al. A randomized, placebo-controlled trial of D-cycloserine for the enhancement of social skills training in autism spectrum disorders. *Molecular autism.* 2016;7:2. doi:10.1186/s13229-015-0062-8
- 33. Hendren RL, James SJ, Widjaja F, Lawton B, Rosenblatt A, Bent S. Randomized, Placebo-Controlled Trial of Methyl B12 for Children with Autism. *Journal of child and adolescent psychopharmacology*. Feb 18 2016;doi:10.1089/cap.2015.0159
- 34. Fujioka T, Inohara K, Okamoto Y, et al. Gazefinder as a clinical supplementary tool for discriminating between autism spectrum disorder and typical development in male adolescents and adults. *Molecular autism*. 2016;7:19. doi:10.1186/s13229-016-0083-y
- 35. Bone D, Bishop S, Black MP, Goodwin MS, Lord C, Narayanan SS. Use of machine learning to improve autism screening and diagnostic instruments: effectiveness, efficiency, and multi-instrument fusion. *Journal of child psychology and psychiatry, and allied disciplines*. Apr 19 2016;doi:10.1111/jcpp.12559
- 36. Guy W. ECDEU Assessment Manual for Psychopharmacology: Publication ADM 76-338. Washington, DC: US Dept of Health, Education, and Welfare. 1976:218-222.
- 37. McCracken JT, McGough J, Shah B, et al. Risperidone in children with autism and serious behavioral problems. *The New England journal of medicine*. Aug 1 2002;347(5):314-21. doi:10.1056/NEJMoa013171
- 38. King BH, Hollander E, Sikich L, et al. Lack of efficacy of citalopram in children with autism spectrum disorders and high levels of repetitive behavior: citalopram ineffective in children with autism. *Archives of general psychiatry*. Jun 2009;66(6):583-90. doi:10.1001/archgenpsychiatry.2009.30
- 39. Bearss K, Johnson C, Smith T, et al. Effect of parent training vs parent education on behavioral problems in children with autism spectrum disorder: a randomized clinical trial. *Jama*. Apr 21 2015;313(15):1524-33. doi:10.1001/jama.2015.3150
- 40. Mazurek MO, Carlson C, Baker-Ericzén M, Butter E, Norris M, Kanne S. Construct Validity of the Autism Impact Measure (AIM). *J Autism Dev Disord*. Jul 2020;50(7):2307-2319. doi:10.1007/s10803-018-3462-8

- 41. Silkey M, Durán-Pacheco G, Johnson M, et al. The Autism Impact Measure (AIM): Meaningful Change Thresholds and Core Symptom Changes Over One Year from an Online Survey in the U.S. *J Autism Dev Disord*. Sep 2023;53(9):3422-3434. doi:10.1007/s10803-022-05635-7
- 42. Wakschlag LS, Briggs-Gowan MJ, Choi SW, et al. Advancing a multidimensional, developmental spectrum approach to preschool disruptive behavior. *J Am Acad Child Adolesc Psychiatry*. Jan 2014;53(1):82-96.e3. doi:10.1016/j.jaac.2013.10.011
- 43. Mazefsky CA, Yu L, White SW, Siegel M, Pilkonis PA. The emotion dysregulation inventory: Psychometric properties and item response theory calibration in an autism spectrum disorder sample. *Autism Res.* Jun 2018;11(6):928-941. doi:10.1002/aur.1947
- 44. Aita SL, Moncrief GG, Greene J, et al. Univariate and Multivariate Base Rates of Score Elevations, Reliable Change, and Inter-Rater Discrepancies in the BRIEF-A Standardization Samples. *Assessment*. Mar 2023;30(2):390-401. doi:10.1177/10731911211055673
- 45. Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. *Sleep*. Dec 15 2000;23(8):1043-51.
- 46. Desai AD, Zhou C, Stanford S, Haaland W, Varni JW, Mangione-Smith RM. Validity and responsiveness of the pediatric quality of life inventory (PedsQL) 4.0 generic core scales in the pediatric inpatient setting. *JAMA Pediatr*. Dec 2014;168(12):1114-21. doi:10.1001/jamapediatrics.2014.1600
- 47. Eapen V, Crnčec R, Walter A, Tay KP. Conceptualisation and development of a quality of life measure for parents of children with autism spectrum disorder. *Autism Res Treat*. 2014;2014;160783. doi:10.1155/2014/160783
- 48. Margolis KG, Buie TM, Turner JB, et al. Development of a Brief Parent-Report Screen for Common Gastrointestinal Disorders in Autism Spectrum Disorder. *J Autism Dev Disord*. Jan 2019;49(1):349-362. doi:10.1007/s10803-018-3767-7
- 49. Taylor L, Gidal B, Blakey G, Tayo B, Morrison G. A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose, Multiple Dose, and Food Effect Trial of the Safety, Tolerability and Pharmacokinetics of Highly Purified Cannabidiol in Healthy Subjects. *CNS Drugs*. Nov 2018;32(11):1053-1067. doi:10.1007/s40263-018-0578-5
- 50. Aran A, Eylon M, Harel M, et al. Lower circulating endocannabinoid levels in children with autism spectrum disorder. *Mol Autism*. 2019;10:2. doi:10.1186/s13229-019-0256-6
- 51. Zou M, Liu Y, Xie S, et al. Alterations of the endocannabinoid system and its therapeutic potential in autism spectrum disorder. *Open Biol.* Feb 2021;11(2):200306. doi:10.1098/rsob.200306
- 52. Voinsky I, Zoabl Y, Shomron N, et al. Blood

RNA sequencing confirms upregulated BATF2 and FCGR1A expression in children

with autism spectrum disorder. <a href="https://www.researchsquare.com/article/rs-1113898/v1">https://www.researchsquare.com/article/rs-1113898/v1</a>; 2021.

- 53. Siani-Rose M, Cox S, Goldstein B, Abrams D, Taylor M, Kurek I. Cannabis-Responsive Biomarkers: A Pharmacometabolomics-Based Application to Evaluate the Impact of Medical Cannabis Treatment on Children with Autism Spectrum Disorder. *Cannabis Cannabinoid Res.* Dec 6 2021;doi:10.1089/can.2021.0129
- 54. Iglesias-Vázquez L, Van Ginkel Riba G, Arija V, Canals J. Composition of Gut Microbiota in Children with Autism Spectrum Disorder: A Systematic Review and Meta-Analysis. *Nutrients*. Mar 17 2020;12(3)doi:10.3390/nu12030792
- 55. Sharon G, Cruz NJ, Kang DW, et al. Human Gut Microbiota from Autism Spectrum Disorder Promote Behavioral Symptoms in Mice. *Cell.* May 30 2019;177(6):1600-1618.e17. doi:10.1016/j.cell.2019.05.004
- 56. Ding X, Xu Y, Zhang X, et al. Gut microbiota changes in patients with autism spectrum disorders. *J Psychiatr Res*. Oct 2020;129:149-159. doi:10.1016/j.jpsychires.2020.06.032